CLINICAL TRIAL: NCT02448238
Title: A Pilot Study of Oral Probiotic Bacteria Supplementation to Reduce Microbial Translocation and Chronic Immune Activation in HIV-infected Malian Women
Brief Title: Pilot Study of Oral Probiotic Bacteria Supplementation to Reduce Chronic Immune Activation in HIV-infected Malian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM15330; VCUHIV001 (Other: VCU)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: HIV
Keywords: Human Immunodeficiency Virus; probiotic; microbial translocation; immune activation; inflammation; VSL#3; Mali; Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- probiotic (Experimental): This is a single arm study all subjects will receive the study VSL#3 probiotic. Subjects will take 1 sachet of powder orally daily for 12 weeks
  Interventions: Other: VSL#3® probiotic

INTERVENTIONS:
Other: VSL#3® probiotic — Other: VSL#3® probiotic VSL#3® DS (Sigma-Tau Pharmaceuticals) is a well characterized water soluble, live (9 × 1011 bacteria/sachet), lyophilized preparation of 8 probiotic bacterium that have been detailed previously. Subjects will take 1 sachet of powder orally daily for 12 weeks. As many Malian homes lack refrigeration, subjects will be issued a special "canari", a commonly used earthenware water container also containing sand that works on the principal of "trans-evaporation" to keep contents at room temperature (~24°C) even in warmer climates. We have verified this in country. Probiotics will be placed in a sealed plastic bag within a sealed jar in the sand of the canari. At the research site, probiotics will be kept refrigerated (4-8°C) in a study provided refrigerator

SUMMARY:
The composition of the intestinal bacterial flora effects gut immunologic function and intestinal barrier integrity. HIV infection impairs gut immune and epithelial function resulting in an altered gut bacterial flora and "leakage" of gut bacterial products into the bloodstream. These bacterial products can overstimulate the immune system leading to increased inflammation and HIV disease progression. The investigators will investigate whether oral supplementation of certain beneficial "probiotic" bacteria may attenuate these processes in HIV infected women in Mali, Africa.

This is a single arm study to evaluate the effect of 12 weeks of combination oral probiotic supplementation (VSL#3, Sigma-Tau Pharmaceuticals - containing 9 × 1011 bacteria of 8 species: S. thermophilus, Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus plantarum, Lactobacillus acidophilus, Lactobacillus paracasei, and Lactobacillus bulgaricus) on plasma biomarkers of immune cell activation, and inflammation. The study population will be 50 chronically HIV-infected but generally healthy, non-pregnant, Malian women subjects with CD4+ T-cell count ≥ 350 cells/mm3 who are not receiving antiretroviral therapy. Blood plasma/serum and fecal sampling will occur at baseline, 4, and 12 week as well as at 24 weeks. At these time points, probiotic will be dispensed, a medical history will be obtained, and adherence will be assessed. Prior to study entry, subjects will have eligibility and safety labs will be obtained and detailed baseline medical and symptom histories, demographics, weight, and stool frequency information will be recorded. A stress assessment questionnaire will be completed at baseline and week 12 to determine the effect of this intervention on stress levels.

The primary study outcome is to assess change (baseline to 12 week) in plasma soluble CD14 (a marker of monocyte response to bacterial endotoxin which has been associated with mortality) with study probiotic. Other outcomes will include assessing change (baseline to 12 week) in plasma interleukin-6, soluble CD163 (another monocyte activation marker), d-dimer (a marker of coagulopathy), intestinal fatty acid binding protein (a marker of gut epithelial cell injury) and fecal calprotectin (a marker of gut inflammation), as well as CD4+ T-cell counts, self reported stool quality (using the Bristol Stool Scale), safety and tolerability of the VSL#3 probiotic, and level of stress.

DETAILED DESCRIPTION:
Excessive immune system stimulation, activation, and associated inflammation play a central role in the pathogenesis of HIV disease. The level of T-cell and monocyte activation predicts the rate of HIV disease progression to AIDS, the slope of CD4+ T-cell loss, and mortality [Liu 1997, Liu 1998, Deeks 2004, Hunt 2008, Sandler 2011]. The mechanism by which HIV disease causes persistent immune activation and inflammation is multifactorial, and includes the direct pathogenic effect of replication, other chronic viral infections, as well as indirect pathways. It is now generally accepted that bacterial translocation into the systemic circulation due to HIV associated gut changes are an important part of this pathology. Both HIV and simian immunodeficiency virus (SIV) infection result in rapid and profound depletion of the gut mucosal Th17+CD4+ T-cells, key immune cells associated with reducing bacterial translocation through the gut wall [Brenchley 2004, Raffetellu 2008]. In addition, both HIV and SIV cause direct damage to intestinal epithelial cells [Li 2008, Nazli 2010], and gene expression studies of the GI mucosa have revealed HIV-associated upregulation of genes involved in inflammatory and apoptotic pathways and downregulation of tight junction [Sankaran 2008]. These HIV-associated gut changes ultimately disrupt the normal synergistic co-existence between man and his/her commensal gut microbial flora, resulting in increased translocation of gut bacterial products such as endotoxin (also known as lipopolysaccharide) and bacterial 16s ribosomal DNA into the systemic circulation. Here, these bacterial products serve as potent stimuli for the sustained T-cell and monocyte activation and inflammation that drive HIV disease progression [Hunt 2008, Brenchley 2006, Jiang 2009]. Treating HIV with antiretroviral therapy (ART) only partially corrects this gut lesion and related inflammatory process.

One possible approach to address this problem is to replenish "ecological niches" in the gut with beneficial bacteria or "probiotics" such as Lactobacillus and Bifidobacillus species, which may be depleted in HIV infected persons and in certain other conditions. Probiotic bacteria and their biofilms have been shown to stimulate innate immunity and result in beneficial metabolic changes that improve gut epithelial barrier and Th17 T-cell functions and reduces gut inflammation and endotoxin leak [Bassaganya-Rievra 2012, Pagnini 2009, Giamarellos-Bourboulis 2009]. This has proven beneficial in several clinical settings including ulcerative colitis, illeal pouch inflammation, and acute diarrhea in children [Tursi 2010, Miele 2009, Minmura 2004, Salari 2012]. In HIV infected individuals, patients treated with ART who fail to attain the expected improvement in blood CD4+ T-cell counts seem to lack the measureable plasma 16s ribosomal DNA signature of Lactobacillus species or have lower fecal concentrations of lactobacillus [Merlini 2011, Perez-Santiago 2013]. Primate SIV models using pigtail macaques have demonstrated that Lactobacillus plantarum supplementation enhances gut Th17 CD4 recruitment, interleukin (IL)-17 expression, epithelial tight junction protein production, and decreases inflammatory chemokines and IL-1B [Sankaran 2013]. Another recent study demonstrated that SIV infected macaques had significantly improved numbers of gut antigen presenting cells and mucosal CD4+ T-cells, reduced gut lymphoid tissue fibrosis, and reduced plasma d-dimer levels when given ART and a combination of probiotic bacteria (VSL#3 and L. rhamnosus CG) vs ART alone [Klatt 2013]. Thus, probiotics could offer important benefits to HIV-infected patients by improving intestinal mucosal and immunologic function and reducing the subsequent bacterial translocation and immune activation that leads to AIDS.

A limited number of studies have looked at probiotics to reduce diarrhea or improve CD4+ T-cell counts in HIV infected individuals, particularly in Africa. Individuals in sub-Sahara Africa are more likely to have diarrhea than in developed countries and the gut microbiome is different [Yatsunenko 2012], as is the greater burden of intestinal parasitosis and pathogenic bacteria such as Salmonella and Cholera. Some data suggest that non-HIV-infected individuals (of African descent as compared to Caucasians, and women as compared with men) may have greater intestinal permeability or display more pronounced systemic inflammatory responses. A study of 24 HIV-infected Nigerian women (CD4+ T-cell count >200, not on ART) with diarrhea were randomized to receive 15 days of yogurt with or without a probiotic (Lactobacillus rhamnosus CG and L. reuteri). The probiotic group had a resolution of diarrhea and stable or improved CD4+ T-cell counts at one month compared to unsupplemented yogurt [Anukam 2008]. Similar CD4 improvements were observed in a randomized probiotic (Bifidobacterium bifidum and Streptococcus thermophilus) study in HIV infected African children [Trois 2008]. An observational study examining the introduction of probiotic yogurt, made by local HIV infected women in a low-income community in Tanzania, was associated with significantly increased CD4+ T-cell counts [Irvine 2010]. Probiotics have proven safe and well tolerated in these and other [Irvine 2011, Kerac 2009, Hummelen 2011, Wolf 1998] studies of HIV infected individuals.

Rationale for Probiotic Bacteria Selection and Safety - All Lactobacillus sp. and other probiotic bacteria may not perform equally well to restore gut mucosal integrity and immune function and do so in a safe fashion. VSL#3® DS (Double-Strength, Sigma-Tau Pharmaceuticals) is a well characterized water soluble, live (9 × 1011 bacteria/sachet, once daily), lyophilized preparation of 8 probiotic bacterium, lacking L. rhamnosus but including previously discussed L. plantarum and S. thermophilus (along with Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus paracasei, and Lactobacillus bulgaricus) that has been studied extensively, with over 140 PubMed citations since 1999. VSL#3 has been shown in vitro and in vivo (rat model) to increase tight junction proteins, reduce intestinal permeability, reduce inflammation, enhance innate immunity, and reduce salmonella invasion [Dai 2012, Mencarelli 2012, Appleyard 2011, Madsen 2001, Pagnini 2010, Gad 2011]. L. paracasei contained within VSL#3 encodes "lactocepin" a protease that selectively degrades secreted and cell-associated chemokines and reduced inflammation in a murine colitis model [von Schillde 2102]. As previously noted, SIV infected macaques had improved numbers of gut antigen presenting cells and mucosal CD4+ T-cells when given VSL#3 and L. rhamnosus vs ART alone [Klatt 2013].

Clinically, VSL#3 has been studied extensively for "pouchitis", which may occur following ileal pouch-anal anastomosis for chronic ulcerative colitis in approximately 30% of patients. Several randomized clinical trial and a Cochrane database review support the safety and efficacy of VSL#3 in reducing acute and chronic pouch inflammation [Holubar 2010]. VSL#3® DS is the only probiotic recognized as an effective tool for the management of pouchitis by the American College of Gastroenterology as well as the German Association of Gastroenterology. Similarly, VSL#3 was an effective adjunct in relapsing mild-to-moderate ulcerative colitis in a double-blind, randomized, placebo-controlled study [Tursi 2010]. In a randomized trial of 59 children with irritable bowel syndrome, VSL#3 was superior to placebo in reducing abdominal pain/discomfort and bloating [Guandalini 2010]. A double-blind, randomized clinical trial of 229 at risk hospitalized patients demonstrated that VSL#3 could prevent antibiotic-associated diarrhea [Selinger 2013]. VSL#3 has been studied in healthy, pregnant Italian women, cirrhotic patients, and critically ill patients with no safety issues [Vitali 2012, Agrwal 2012, Gupta N 2013, Frohmader 2010].

As previously noted, the medical literature identifies only rare cases of lactobacillus or bifidobacillus bacteremia (not associated with VSL#3), generally in severely immune compromised patients or nosocomial, central line associated infections on persons not taking probiotic. An 8 year retrospective study in a large U.S. academic medical center found a maximum 0.2% probiotic bacteremia incidence among hospitalized probiotic recipients [Simkins 2013]. An extensive review by the U.S. Department of Health and Human Services (DHHS) completed in 2011 of 387 case series and randomized controlled trials involving over 24,000 patients found no cases where use of a product including Lactobacillus, Bifidobacterium, Saccharomyces, Streptococcus, Enterococcus, or Bacillus led to a hospital admission [Hempel 2011]. Evidence for hospital admissions or bacteremias due to probiotics use came only from case reports and were rare. The DHHS study found no evidence of increased adverse effects associated with probiotic use but added that "rare adverse events are difficult to assess, and despite the substantial number of publications, the current literature is not well equipped to answer questions on the safety of probiotic interventions with confidence". An independent panel of food safety experts concluded that VSL#3® is "Generally Recognized As Safe (GRAS) for medical food use." GRAS is an U.S. Food and Drug Administration (FDA) designation that acknowledges certain food additives as safe under the conditions of their intended use by qualified experts. To receive such recognition, the product must establish a consensus of expert opinion regarding the safety of its use based on a review of scientific evidence.

Rationale for a Single Arm Design - The hypothesis being tested is that oral probiotic bacteria supplementation will reduce endotoxemia and endotoxin-associated macrophage and T-cell activation in HIV-infected subjects. Because we expect endotoxin and macrophage/T-cell activation levels to remain stable (or perhaps slowly increase) in subjects who are not receiving ART [Deeks 2004], a single arm study will allow us to determine whether the intervention has an effect. In this study, individuals with CD4+ T-cell counts >350 cells/mm3 will be enrolled. Among persons with CD4+ T-cell counts >350 cells/mm3, the rate of AIDS and non-AIDS events was 0.7 events per 100 person-years [Baker 2008], so investigators expect these complications to be unlikely during the study. Recently, WHO guidelines have changed to recommend starting ART when the HIV infected individual's CD4+ T-cell counts is <500 cells/mm3 so it is likely that some subjects would now be recommended for ART. However, ART availability is currently limited in this region so many potential subjects could participate until such time as ART is more broadly available. Subjects with plans to initiate ART within the study duration of 24 weeks will not be enrolled.

STUDY DESIGN - This is a single arm study to evaluate the effect of 12 weeks of combination oral probiotic supplementation (VSL#3) on biomarkers of microbial translocation, monocyte and T-cell activation, and inflammation in the blood in chronically HIV-infected Malian women subjects with CD4+ T-cell count ≥ 350 cells/mm3 who are not receiving ART. Subjects will be re-evaluated at week 24 to determine sustainability of any changes. This study will enroll 50 subjects. Blood plasma/serum and fecal sampling will occur at baseline, 4, 12, and 24 weeks. All subjects will be examined for intestinal parasites within 45 days before study entry. Detailed demographic, weight and BMI, stool frequency, symptoms, ART history, CD4 and HIV RNA will be recorded. A stress assessment questionnaire will be completed at baseline and week 12

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, or plasma HIV-1 RNA viral load.
* No plans to initiate ART during the course of the proposed study. NOTE: Subjects who meet WHO treatment guidelines for initiating ART once enrolled should begin therapy as clinically indicated. These subjects must stop study treatment, and will be followed on study/off study treatment.
* Screening CD4+ T-cell count ≥ 350 cells/mm3 performed in a laboratory that has a Malian National Institute for Public Health and Research (INRSP) certification, or its equivalent, within 45 days prior to study entry.
* Laboratory values obtained within 45 days prior to entry as follows:

  * Absolute neutrophil count (ANC) ≥ 1000/mm3
  * Hemoglobin ≥ 10.0 g/dL
  * Platelet count ≥ 50,000/mm3
* Female subjects of reproductive potential [defined as girls who have reached menarche or women who have not been post-menopausal for at least 12 consecutive months, i.e., who have had menses within the preceding 12 months, or have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or bilateral tubal ligation)] must have a negative serum or urine pregnancy test performed within 45 days prior to entry.
* Female subjects participating in sexual activity that could lead to pregnancy must agree to use at least one of the following forms of birth control for at least 45 days prior to study entry until the final study visit:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive (pill, injection, implants)
* Female subjects who are not of reproductive potential are eligible without requiring the use of a contraceptive. Acceptable documentation of sterilization, other contraception methods, menopause and reproductive potential is patient-reported history at any time prior to or during screening.
* Malian women age => 18 years.
* Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

* Pregnant.
* Use of any antiretroviral agent during or within 24 weeks prior to study entry.
* Use of any of the following medications for more than 3 consecutive days during or within 45 days prior to study entry:

  * Immunosuppressives
  * Immune modulators
  * Antineoplastic/Anticancer agents
  * Probiotics
  * Anticoagulants ( Aspirin is permitted )
* Known allergy/sensitivity/intolerance to any probiotic formulation. Lactose intolerance is not exclusionary unless there was a hypersensitivity reaction
* Active illicit drug or alcohol use or dependence, or conditions that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness or trauma requiring systemic treatment and/or hospitalization within 45 days prior to study entry. Chronic stable conditions such as hypertension or diabetes are not exclusionary.
* Anticipated antibiotic use during the study or use within 45 days prior to study entry. Topical antibiotics are permitted.
* Known cirrhosis or severe liver disease (e.g., ascites, encephalopathy, history of variceal bleeding).
* Recent (within 12 weeks) history of, or active, bowel obstruction, inflammatory bowel disease, colitis, intestinal bleeding, GI malignancy, or severe GI motility disorders including severe constipation or severe diarrhea (>5 stools day/average) or severe swallowing disorders.
* Active gastrointestinal parasitic infection.
* Major GI tract surgery within 45 days prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
change in plasma soluble CD14 (sCD14) | baseline to week 12
  sCD14 is marker of monocyte response to endotoxin associated with mortality

SECONDARY OUTCOMES:
change in plasma soluble CD163 (sCD163) | baseline to week 12
  sCD163 is a marker of monocyte activation associated with cardiovascular disease (CVD)
change in plasma interleukin-6 (IL-6) | baseline to week 12
  IL-6 is associated with mortality and CVD
change in plasma d-dimer | baseline to week 12
  d-dimer is associated with mortality and CVD
change in plasma intestinal fatty acid biding protein | baseline to week 12
  intestinal fatty acid biding protein is associated with gut epithelial cell injury
change in CD4+ T cell counts | baseline to week 12
  CD4 is associated with HIV disease progression
change in fecal calprotectin | baseline to week 12
  fecal calprotectin is associated with gut inflammation
change in stress levels | baseline to week 12
  uses standardized questionnaire
number of participants with NIH/Department of AIDS Grade ≥ 2 signs and symptoms, Grade ≥ 2 laboratory abnormalities and other serious adverse events | baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Nixon, DO, PhD, Principal Investigator — Virginia Commonwealth University, USA; Saba Masho, MD, MPH, Study Director — Virginia Commonwealth University, USA; Susan Kornstein, MD, Study Director — Virginia Commonwealth University, USA
Locations (1):
- Nianankoro Fomba Hospital, Ségou, Ségou, Mali